CLINICAL TRIAL: NCT02012218
Title: A Phase 3b, Multicenter, Open-label Exploratory Trial to Evaluate the Efficacy, Safety, and Subject Satisfaction With Brexpiprazole as Adjunctive Therapy in the Treatment of Adults With Major Depressive Disorder and an Inadequate Response to Previous Adjunctive Therapy
Brief Title: Brexpiprazole as Adjunctive Therapy With Major Depressive Disorder and an Inadequate Response to Previous Adjunctive Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-13-001
Record Dates: First submitted 2013-12-04; First posted 2013-12-16 (Estimated); Results first posted 2015-10-08 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder, Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADT and Brexpiprazole (Experimental): ADT and Brexpiprazole
  Interventions: Drug: ADT; Drug: Brexpiprazole

INTERVENTIONS:
Drug: ADT
Drug: Brexpiprazole

SUMMARY:
The objectives of this exploratory trial are to evaluate the efficacy, safety, and subjects' subjective satisfaction when switching to adjunctive brexpiprazole in subjects with MDD who have responded inadequately to preceding adjunctive drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MDD
* In current major depressive episode of ≥ 8 weeks in duration and includes an inadequate response to at least 1 adjunctive treatment.
* Positive history of at least 1 additional failure to an adequate monotherapy antidepressant treatment.
* HAM-D17 total score≥ 18
* Currently receiving SSRI of SNRI with adjunctive treatment for at least 6 weeks before screening.
* Willing to discontinue use of all prohibited psychotropic medications
* Historical positive serological results for HIV, hepatitis B/C
* Able to provide written informed consent prior to the initiation of any protocol-required procedures
* Subjects who could potentially benefit from adjunctive treatment with Brexpiprazole

Exclusion Criteria:

* Sexually active women of childbearing potential
* Male subjects not practicing 2 different methods of birth control
* Females who are breastfeeding and/or who have a positive pregnancy test result
* Subjects who have received ECT for the current major depressive episode.
* Subjects who have had an inadequate response to ECT
* Current need for involuntary commitment or who have been hospitalized within 4 weeks of screening
* Current Axis I (DSM-IV-TR)
* Current Axis II (DSM-IV-TR)
* Subjects experiencing hallucinations, delusions, or any psychotic symptomatology in the current major depressive episode.
* Subjects receiving new onset psychotherapy.
* Subjects who answer "Yes" on the C-SSRS Suicidal Ideation Item 4, Item 5, or on any of the 5 C-SSRS Suicidal Behavior Items
* Subjects who have met DSM-IV-TR criteria for substance abuse or dependence within the past 180 days
* Hypothyroidism or hyperthyroidism
* Clinically significant neurological, hepatic, renal, metabolic, haematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders
* Currently treated with insulin for diabetes
* Uncontrolled hypertension or symptomatic hypotension, or orthostatic hypotension
* Known ischemic heart disease or history of myocardial infarction, congestive heart failure, angioplasty, stenting, or coronary artery bypass surgery
* Epilepsy or history of seizures
* Positive drug screen
* The following laboratory test and ECG results are exclusionary:

  1. Platelets ≤ 75,000/mm3
  2. Hemoglobin ≤ 9 g/dL
  3. Neutrophils, absolute ≤ 1000/mm3
  4. AST > 2 × ULN
  5. ALT > 2 × ULN
  6. CPK > 3 × ULN, unless discussed with and approved by the medical monitor
  7. Creatinine ≥ 2 mg/dL
  8. HbA1c ≥ 7.0%
  9. Abnormal free T4 (Note: Free T4 is measured only if result for TSH is abnormal.)
  10. QTcF ≥ 470 msec for females and ≥ 450 msec for males
* Treatment with an MAOI or EMSAM within 14 days of the Baseline visit.
* Use of benzodiazepines and/or hypnotics within 7 days prior to the first dose of IMP
* Use of oral neuroleptics within 7 days prior or long-acting approved atypical antipsychotics ≤ 1 full cycle plus ½ cycle prior to the first dose of IMP
* Subjects who would be likely to require prohibited concomitant therapy during the trial.
* Subjects who previously participated in any prior brexpiprazole trial
* History of neuroleptic malignant syndrome or serotonin syndrome
* History of true allergic response to more than one class of medications
* Prisoners or subjects who are compulsorily detained for treatment of either a psychiatric or physical illness.
* Subjects who participated in a clinical trial within the last 180 days or who participated in more than 2 clinical trials within the past year.
* Any subject who, in the opinion of the investigator or medical monitor, should not participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd Japan (OPCJ)
Locations (24):
- United States (24):
  - Collaborative NeuroScience Network, Inc., Garden Grove, California
  - Viking Clinical Research, Ltd., Temecula, California
  - Clinical Neuroscience Solutions Pharmacology, Orlando, Florida
  - Carman Research, Smyrna, Georgia
  - Goldpoint Clinical Research, Indianapolis, Indiana
  - Alpine Clinic, Lafayette, Indiana
  - Pharmasite Research, Baltimore, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Coastal Research Associates, Inc., Weymouth, Massachusetts
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - St. Louis Clinical Trials, St Louis, Missouri
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Behavioral Medical Research of Staten Island, Staten Island, New York
  - Richard H. Weisler, MD, PA, Raleigh, North Carolina
  - Midwest Clinical Research Center MCRC, Dayton, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Lincoln Research, LLC, Lincoln, Rhode Island
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Future Search Trials of Dallas, LP, Dallas, Texas
  - NeuropsychiatricAssociates, Woodstock, Vermont
  - Frontier Institute, Spokane, Washington

REFERENCES:
- [Derived] Weiss C, Meehan SR, Brown TM, Gupta C, Morup MF, Thase ME, McIntyre RS, Ismail Z. Effects of adjunctive brexpiprazole on calmness and life engagement in major depressive disorder: post hoc analysis of patient-reported outcomes from clinical trial exit interviews. J Patient Rep Outcomes. 2021 Dec 11;5(1):128. doi: 10.1186/s41687-021-00380-4. PMID 34894307
- [Derived] Fava M, Okame T, Matsushima Y, Perry P, Weiller E, Baker RA. Switching from Inadequate Adjunctive or Combination Treatment Options to Brexpiprazole Adjunctive to Antidepressant: An Open-Label Study on the Effects on Depressive Symptoms and Cognitive and Physical Functioning. Int J Neuropsychopharmacol. 2017 Jan 1;20(1):22-30. doi: 10.1093/ijnp/pyw087. PMID 27784751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted in 61 participants in 28 trial sites, all of which were located in the United States.
Pre-assignment Details: The trial consisted of a continuous 6-week open-label treatment period including an initial 2-week titration period with a 30-day (+2 days) follow-up period.
Groups:
- Group 1A: Participants who had received a prescribed number of tablets of aripiprazole (baseline/primary antidepressant therapy [ADT]) and adjunctive therapy were switched to ADT plus one tablet of brexpiprazole as adjunctive therapy daily throughout the 6-week treatment period.
- Group 1B: Participants who had received a prescribed number of tablets of quetiapine IR (immediate release) or XR (extended release) (baseline/primary ADT) and adjunctive therapy were switched to ADT plus one tablet of brexpiprazole as adjunctive therapy daily throughout the 6-week treatment period.
- Group 2: Participants who had received a prescribed number of tablets of any Selective Serotonin Reuptake Inhibitors (SSRI), any Serotonin-norepinephrine Reuptake Inhibitors (SNRI), any tricyclic antidepressant, or Oleptro (trazodone hydrochloride) IR or XR (baseline/primary ADT) and adjunctive therapy were switched to ADT plus one tablet of brexpiprazole as adjunctive therapy daily throughout the 6-week treatment period.
- Group 3: Participants who had received a prescribed number of tablets of bupropion (baseline/primary ADT) and adjunctive therapy were switched to ADT plus one tablet of brexpiprazole as adjunctive therapy daily throughout the 6-week treatment period.
- Group 4: Participants who had received a prescribed number of tablets of stimulants such as modafinil, methylphenidate, or psychostimulant (baseline/primary ADT) and adjunctive therapy were switched to ADT plus one tablet of brexpiprazole as adjunctive therapy daily throughout the 6-week treatment period.
Period: Overall Study
Arm/Group | Group 1A | Group 1B | Group 2 | Group 3 | Group 4
Started | 12 | 11 | 13 | 19 | 6
Completed | 8 | 10 | 11 | 17 | 5
Not Completed | 4 | 1 | 2 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0
Not completed — Protocol Specified | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1A | Group 1B | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 12 | 11 | 13 | 19 | 6 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.2 (8.13) | 41.8 (13.57) | 48.5 (12.20) | 44.1 (13.64) | 41.7 (13.59) | 45.6 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 11 | 15 | 3 | 43
  Male | 5 | 4 | 2 | 4 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 6 in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS was used as the primary efficacy assessment of level of depression. The MADRS was administered using the Structured Interview Guide for the MADRS. Detailed instructions were provided.The MADRS consists of 10 items each, with 7 defined grades of severity (ie, 0 to 6, with 0 being the "best" rating and 6 being the "worst" rating). The MADRS total score is the sum of ratings for all 10 items; therefore, possible total scores range from 0 to 60. The MADRS total score least squares (LS) mean changes from baseline to Week 6 is mentioned below.
Time Frame: Baseline and Week 6
Population: All participants who took at least one dose of brexpiprazole and who had a valid baseline assessment and at least one valid post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Group 1A | Group 1B | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 12 | 10 | 12 | 19 | 6
Units on a scale | -12.8 (2.26) | -18.4 (2.10) | -19.5 (1.99) | -19.2 (1.59) | -16.8 (2.97)
Statistical Analysis 1: Comparison: Group 1A vs Group 1B vs Group 2 vs Group 3 vs Group 4; The null hypothesis of zero in mean change from baseline in MADRS total score at Week 6 was tested for each treatment group at significance level of 0.05 (2-sided); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis — P-values were calculated according to testing a null hypothesis of zero mean change; This analysis was conducted using a mixed model repeated measures analysis on observed case data

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent until the end of trial with a safety follow-up of 30 (+2 ) days.
Arm/Group | Group 1A | Group 1B | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/11 | 0/13 | 0/19 | 0/6
Other Adverse Events (participants affected / at risk) | 7/12 | 8/11 | 6/13 | 15/19 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1A (N=12) | Group 1B (N=11) | Group 2 (N=13) | Group 3 (N=19) | Group 4 (N=6)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1A (N=12) | Group 1B (N=11) | Group 2 (N=13) | Group 3 (N=19) | Group 4 (N=6)
Akathisia (Nervous system disorders) | 2 | 0 | 0 | 3 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 2 | 1
Disturbance in attention (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 2 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Glabellar reflex abnormal (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Disinhibition (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Distractibility (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Middle insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 1 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 2 | 3 | 3
Increased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 2 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Food craving (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Menstrual disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No